CLINICAL TRIAL: NCT06034834
Title: Near-Infrared Imaging for Perfusion Assessment of Traumatic Soft Tissue and Skeletal Injuries
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Joost R. van der Vorst, MD, PhD, Dr. J. R. van der vorst, Vascular Surgeon, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL84014.058.23
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Perfusion; Traumatic Injury; Fluorescence Imaging
Keywords: Indocyanine Green; Near-infrared fluorescence imaging; Traumatic injuries; Perfusion
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The study is a prospective observational multicentre pilot study. All included patients will undergo a perfusion assessment using ICG NIR fluorescence imaging. Perfusion assessment will not affect the treatment of patients.
Masking Description: The surgeons will be blinded as to the results of the intraoperative perfusion assessment in order to prevent bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traumatic injuries (Experimental): Acute patients treated surgically for:
  * Open deglovement (n=20)
  * Crush injury (n=20)
  * Open fractures (n=20)
  The setting is defined acute when there is less than 24 hours between sustaining the injury and surgery.
  Elective patients treated surgically for:
  * Fracture related infection (FRI) (n=10)
  * Non-union of fractures (n=50) Subdivided into 5 groups of 10.
    * Elective osteosynthesis of non-union clavicula fracture N=10
      * Primarily operated on N=5
      * Primarily treated conservatively N=5
    * Elective osteosynthesis of non-union tibia. N=10
    * Elective osteosynthesis of non-union ulna. N=10
      * Primarily operated on N=5
      * Primarily treated conservatively N=5
    * Elective osteosynthesis of non-union humerus. N=10
    * Elective osteosynthesis of non-union of the rib. N=10
  Interventions: Diagnostic Test: Near-infrared fluorescence imaging of perfusion

INTERVENTIONS:
Diagnostic Test: Near-infrared fluorescence imaging of perfusion — Patients will undergo an intra-operative perfusion assessment using ICG NIR fluorescence imaging after clinical judgment and debridement of the traumatic injury. For patients undergoing additional debridement procedures, perfusion assessment with ICG will be repeated during every procedure.

SUMMARY:
To date, intraoperative assessment of tissue and bone viability is predominantly subjective, depending on the clinical view of the surgeon, resulting in a variation in the thoroughness of debridement. Inadequate initial resection leads to multiple debridement interventions, leading to prolonged hospitalization or readmission with consequently high direct medical costs.

Near-Infrared Fluorescence (NIRF) imaging with Indocyanine Green (ICG) could potentially be a relevant contribution to adequately treating soft tissue and skeletal injuries by creating an improved distinction between viable and non-viable tissue, based on perfusion indices.

This study evaluates whether intraoperative perfusion assessment with ICG fluorescence imaging is a feasible and quantifiable technique for treating traumatic injuries.

DETAILED DESCRIPTION:
Rationale: In 2020 71.623 Dutch patients were acutely admitted to hospitals due to sustained traumatic injuries. 7% of the injuries related to open wounds and 44% to fractures. The majority of traumatic musculoskeletal injuries needs to be diagnosed and treated as soon as possible to lower the risk of infections and to minimize adverse outcome, such as necrosis and/or osteomyelitis. To date, intraoperative assessment of tissue and bone viability is predominantly subjective, resulting in a variation in thoroughness of debridement. If not all necrotic tissue is removed, suboptimal healing occurs, which serves as a potential food source for bacteria. In addition, inadequate initial resection leads to multiple debridement interventions, leading to prolonged hospitalization or readmission with consequently high direct medical costs. Since tissue necrosis is an ongoing process, radical resection of avital tissue during the initial procedure is not always possible. The surgeon's visual estimation is not optimal to predict the final amount of debridement. After maximal debridement, antibiotic treatment and coverage of open wounds, the incidence of infection can rise to 27%. Compromised perfusion is at the centre of this problem. An adequate blood supply is crucial for tissue viability and infection clearance.

Near-Infrared Fluorescence (NIRF) imaging with Indocyanine Green (ICG) has already shown its potential in effective real-time assessment of intra-operative tissue perfusion and the early prediction of future necrosis in multiple studies. This technique could potentially be a relevant contribution in adequately treating soft tissue and skeletal injuries by creating an improved distinction between viable and non-viable tissue, based on perfusion indices. However to date, the feasibility to quantify this technique in posttraumatic tissue has not been successfully evaluated.

Objective: The primary objective of this study is to evaluate the feasibility of Near-infrared Fluorescence (NIRF) imaging with Indocyanine green (ICG) to assess and quantify tissue perfusion in post-traumatic soft tissue and/or skeletal injury.

Study design: The study is a prospective observational multicentre pilot study. All included patients will undergo a perfusion assessment using ICG NIR fluorescence imaging. Perfusion assessment will not affect treatment of patients.

Study population: Patients aged 18 years or older with traumatic soft tissue and/or skeletal injury. Injuries included in the study are: open deglovement; crush injuries of extremities; open fractures, non-unions of clavicula, tibia, humerus, rib and/or ulna fractures and fracture related infections.

Intervention: Patients will undergo an intra-operative perfusion assessment using ICG NIR fluorescence imaging. For patients undergoing additional debridement procedures, perfusion assessment with ICG will be repeated during every procedure.

Main study parameters/endpoints: The primary outcome of this study is a time-intensity curve with quantified perfusion parameters in traumatic soft tissue and/or skeletal injuries. Perfusion parameters included in the analyses are time till maximum intensity (Tmax), maximum intensity (Imax) the ingress rate, the normalized slope, the absolute slope and the area under the curve at 30, 60 and 120 seconds.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all the following criteria:

* Age ≥ 18 years
* Diagnosed with one or more of the following injuries:

  * Crush injury
  * Open deglovement
  * Open fracture(s) (Gustilo 3, -A, -B & -C)
  * Non-union tibia/clavicula/ulna/humerus/rib
  * Fracture related infection
* Indication for surgical intervention

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Hemodynamically unstable due to severe blood loss
* Allergic or hypersensitive to iodine/crustaceans/shellfish
* Diagnosed with endocrine thyroid disorders (hyperthyroidism)
* Pregnancy
* Diagnosed with impaired renal function eGFR <30 L/min/1.73m2
* Diagnosed with severely disturbed hepatic enzymes/liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Time-intensity curves | 1 day
  The main endpoint of this study is an adequate time-intensity curve extracted from selected regions of interest. Adequate curves are defined as reproducible curves with accurate representation of the perfusion status. An adequate curve is characterized by a recognisable in- and outflow pattern representing the bloodflow in the tissue. Distinguishing between adequate, questionable and inadequate perfusion can only be done after comparing the measurement results.

SECONDARY OUTCOMES:
Maximum intensity (Imax) | 1 day
  As secondary study parameters quantified perfusion parameters will be extracted from the time-intensity curves. The parameters extracted include:
  • Maximum intensity (Imax) in arbitrary units (a.u.)
Time till maximum intensity (Tmax) | 1 day
  As secondary study parameters quantified perfusion parameters will be extracted from the time-intensity curves. The parameters extracted include:
  • Time till maximum intensity (Tmax), in seconds.
The ingress rate and absolute slope | 1 day
  As secondary study parameters quantified perfusion parameters will be extracted from the time-intensity curves. The parameters extracted include:
  * The ingress rate
  * The absolute slope Both in arbitrary units per second (a.u./s)
The normalized slope | 1 day
  As secondary study parameters quantified perfusion parameters will be extracted from the time-intensity curves. The parameters extracted include:
  • The normalized slope in percentages per second (%/s)
The area's under the curve at 30, 60 and 120 seconds | 1 day
  As secondary study parameters quantified perfusion parameters will be extracted from the time-intensity curves. The parameters extracted include:
  • Area under the curve at 30, 60 and 120 seconds in percentages (%)
Incidence of necrotic tissue | 90 days of necrotic
  Perfusion parameters will be evaluated for their correlation with the occurrence of necrotic tissue after initial debridement.
  This will be calculated as the percentage of people with inadequate perfusion parameters that develop necrotic tissue compared to people with adequate perfused tissue.
The amount of additional debridement procedures | 90 days
  The number of additional debridement procedures when comparing the group with inadequate perfused tissue to the group with adequate perfused tissue.
  In numbers and percentages.
The infection incidence | 90 days
  Perfusion parameters will be evaluated for their correlation with the occurrence of wound infection within 90 days after procedure. Infection defined as a red, swollen and painful area that is warm and tender to touch, possibly in combination with fever/chills, purulent effusion, positive cultures or increased infection parameters. The group with adequate perfused tissue will be compared to the group with inadequate perfusion.
  This will be in numbers and percentages.
The incidence of a fracture related infection | 90 days
  Incidence of a fracture related infection will be compared between the groups with adequate and inadequate perfusion in numbers and percentages.
Lentgh of hospital stay | 90 days
  The length of hospital stay will be measured in days and compared between groups with adequate and inadequate perfusion.
Amount of readmission | 90 days
  The number of readmissions within 90 days associated with complications of primary problem (infection, necrosis, death) will be compared between the groups with inadequate and adequate tissue perfusion in numbers and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Koning, MD, Study Director — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus University Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No